CLINICAL TRIAL: NCT04271007
Title: Phase IV Clinical Study,Comparative, Blind Double and Randomized to Compare Mometasone Furoate Cream (TOPISON) Versus Other Two Cream Mometasone Furoate, in Participants With Atopic Dermatitis
Brief Title: Comparative Study:Topison (Mometasone Furoate) Versus Two Others Mometasone Furoates
Acronym: LB2001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EN19092501
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2022-07

CONDITIONS: Atopic Dermatitis
Keywords: Topison; Atopic dermatitis; mometasone furoate
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Mometasone Furoate

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups, as follows:
  Group I: Use the drug Topison on one side of the upper limb and Mometasone Furoate 1mg /g Sanofi,Medley on the opposite side.
  Group II: Use the drug Topison on one side of the upper limb and Mometasone Furoate 1mg / g Ache on the opposite side.
  The side of the upper limb for the use of Topison or momofasone furoate Sanofi,Medley or Aché will be defined randomly.
Who Masked: Participant, Investigator
Masking Description: To allow the study to be blinded, each participant will receive the product from the non-blind professional, delegated by the Principal Investigator, according to the allocation generated through the randomization list. Uncharacterized products will be dispensed with, making it impossible to identify them. The cream that each participant will receive will be non-transferable and confidential to the other research participants and to the employees of the research center, except for the non-blind professional; therefore, the research center should guide this conduct when dispensing.
  The Sponsor will delegate a non-blind monitor other than the monitors responsible for the study's monitoring. The non-blind monitor will be responsible only for checking the randomization, accounting and adherence of the returned medication. This conference should be held in a room isolated from the other monitors in the study and other professionals in the research center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Use of the drug Topison on one side of the upper limb and Mometasone Furoate 1mg /g Sanofi, Medley on the opposite side
  Interventions: Drug: Mometasone Furoate
- Group II (Active Comparator): Use of the drug Topison on one side of the upper limb and Mometasone Furoate 1mg /g Aché on the opposite side
  Interventions: Drug: Mometasone Furoate

INTERVENTIONS:
Drug: Mometasone Furoate — mometasone furoate

SUMMARY:
Atopic dermatitis is a chronic disease, with outbreaks, predominant in childhood, whose main symptom is pruritus of variable intensity and signs of cutaneous xerosis and eczematous pattern lesions.

In this context, the present study aims to evaluate a comparative way of Topison drugs in reducing transepidermal water loss, improving skin hydration and comfort in participants with atopic dermatitis.

DETAILED DESCRIPTION:
Phase IV, national, single-center, comparative, double-blind, randomized clinical study with instrumental, clinical and subjective tests to compare mometasone cream puncture (Topison) versus two other mometasone cream punctures in participants with atopic dermatitis.

60 research participants of both sexes will be required, aged 10 or over and under or equal to 60 years.

Participants will be randomized into two groups, as follows:

Group I: Use the drug Topison on one side of the upper limb and Mometasone Furoate 1mg / g Sanofi, Medley on the opposite side.

Group II: Use the drug Topison on one side of the upper limb and Mometasone Furoate 1mg / g Aché on the opposite side.

The side of the upper limb for the use of Topison or momofasone furoate Sanofi, Medley or Aché will be defined randomly.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and consent / consent to their participation in this clinical study, manifested by signing the Informed Consent Form and, when applicable, the Informed Consent Form and the responsible consent form;
* Participants of both sexes aged 10 or over and less than or equal to 60 years;
* Participant with a previous history of atopic dermatitis (who has had at least one crisis in his life);
* Presence of active lesions of atopic dermatitis in the upper limbs in a symmetrical way that allows the treatment of two different regions with two different products. Both lesions must be present with the following symptoms: dry skin, itching and erythema with mild (1) or moderate (2) intensity, assessed using the scale: 0: absent, 1: mild; 2: moderate and 3: intense;
* Agreement to follow the trial procedures and attend the clinic on certain days and times.

Exclusion Criteria:

* Pregnancy / lactation or intention to record during the study period;
* Women who do not agree to use acceptable contraceptive methods (oral contraceptive, injectable contraceptive, intrauterine device (IUD), hormonal implant, barrier methods, hormonal transdermal patch and tubal ligation); except for those that are surgically sterile (bilateral oophorectomy or hysterectomy), as menopausal women for at least 01 (one) year and as participants who declared that they did not practice sexual practices or exercise in a non-reproductive manner;
* Male participants who do not agree to use acceptable contraceptive methods:

Contraceptive methods for the participant: barrier condom, except for those who are surgically sterile (vasectomy) or for a participant in sexual abstinence; Contraceptive methods for partner: oral contraceptive, injectable contraceptive, intrauterine device (IUD), hormonal implant, hormonal transdermal patch, tubal ligation and pressure inhibition methods for women who are sterile (bilateral oophorectomy or hysterectomy), menopausal at least 01 (one) year;

* Use of the following medications for topical or systemic use: antihistamines, non-hormonal anti-inflammatory drugs, antibacterial, antifungal and corticoid with no period less than or equal to 30 days before the selection data;
* Participants with fungal and / or bacterial infections at the time of selection;
* Decompensated endocrinopathies;
* Relevant or current medical history of alcohol or other drug abuse;
* Known history or suspected intolerance / allergy to products of the same category or components of the formula;
* Intense sun exposure up to 15 days before the evaluation;
* Aesthetic or dermatological treatment in the evaluation area up to 4 weeks before selection;
* Professionals directly involved in carrying out the present study;
* Other conditions of use by the evaluating physician as reasonable to disqualify participation in the study. If so, it can be described under observation in the clinical record.
* Use of the following medications for topical or systemic use: antihistamines, non-inflammatory drugshormonal, antibacterial, antifungal, immunosuppressive and corticosteroids in the period less than or equal to 30 daysbefore the date of selection.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
sensory evaluation | up to 5 minutes after first monitored aplication
  Compare performance in the immediate burning sensation after the first monitored application, assessed by the research participant through sensory evaluations
Effectiveness | after 15 days of using the products.
  Compare the effectiveness of Topison cream and two other Mometasone Furoate products in reducing transepidermal water loss by Evaporimetry (TEWL) after 15 days of using the products.

SECONDARY OUTCOMES:
Hydrating efficacy using the equipment Corneometer MPA 580 (Courage Khazaka) | after 15 days of use using instrumental measures
  Compare the hydrating efficacy of Topison cream medications and two other Mometaona Furoate products after 15 days of use using instrumental measures by the Corneometer® equipment.Corneometer equipment measures skin hydration by capacitance. A device probe is a capacitor that, during a measurement, forms an electric field that is interfered by the water present in the skin. The device displays the amount of water present in the arbitrary units, intrinsic to the equipment, from 0 to 130. Without changes, a probe / capacitor interprets the result as 0 and, when affected by the water present on the skin, it presents higher results. The greater the amount of water present on the skin, the higher the result of the application, therefore, it is expected that the values will increase after the application of the product.
Sensory parameters (immediate burning, spreadability, feeling of comfort and calming effect) | after 15 days of continuous use.
  Compare the performance of Topison cream and two other Mometasone Furoate products through sensory parameters, evaluated by the research participant after the first monitored application and after 15 days of continuous use.The participant will evaluate:
  Regarding the immediate burning sensation after applying the product, the alternative applicable to what was felt:Intense, moderate, light, very light, absent (without burning).About product spreadability:very difficult (impossible to spread),spreadability difficult, normal, easy, spreadability very easy (pleasant) If the product provides a comfortable feeling for the skin: strongly disagree, disagree, I do not agree nor disagree,accept,I fully agree. And finally, if the product provides a calming effect for your skin: completely disagree, disagree, neither agree nor disagree, agree, fully agree.
Improvement in atopic dermatitis symptoms:erythema, edema, excoriation, crust, lichenification, dry skin and pruritus | after 15 days of continuous use
  Compare the improvement in atopic dermatitis symptoms between Topison cream and two other Mometasone Furoate products after 15 days of continuous use, compared to baseline thorugh clinical evaluation performed by dermatologist.The dermatologist will evaluate the signs and symptoms: erythema, edema, abrasion, crust, lichenification, dry skin and itching according to an intensity scale: absent (0), mild (1), moderate (2) and this scale (zero) represents the best result and 3 the worst.
Improvement in atopic dermatitis symptoms (questionnaire) | after 15 days of continuous use
  Compare the improvement in atopic dermatitis symptoms between Topison cream and two other Mometasone Furoate products after 15 days of continuous use, using a questionnaire evaluated by the research participant.The participant will answer two questions in this questionnaire:
  1. hydration status of your skin after using the product
  2. If the product reduces any itchy sensations on the skin.
  The answer options for both questions will be:
  it got worse, it didn't change, it improved little, it improved modernly or it improved (following a descriptive scale from the worst scenario to the best).
Preference assessment | after 15 days of continuous use
  Assess which product the research participant prefers, among the two he has used, after 15 days of continuous use.The subject will inform if the best product was applied to the right or left arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Sérgio Sckalka, Osasco, São Paulo, Brazil